CLINICAL TRIAL: NCT02549794
Title: Comparison of Image Quality of Coronary Computed Tomography Angiography bEtweeN High concenTRATion and Low concEntration Contrast Agents(CONCENTRATE Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 4-2015-0173
Record Dates: First submitted 2015-08-16; First posted 2015-09-15 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: low concentration contrast agent; Low dose contrast agent; computed tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High concentration (370) (Active Comparator): CT angiography with hign concentration iodine contrast agent of 370 mg iodine/ml
  Interventions: Procedure: CT angiography with high concentration contrast agent
- Low concentration (320) (Experimental): CT angiography with low concentration iodine contrast agent of 320 mg iodine/ml
  Interventions: Procedure: CT angiography with low concentration contrast agent (320)
- Low concentration (270) (Experimental): CT angiography with low concentration iodine contrast agent of 270 mg iodine/ml
  Interventions: Procedure: CT angiography with low concentration contrast agent (270)

INTERVENTIONS:
Procedure: CT angiography with high concentration contrast agent — Standard concentration of iodine contrast agent for CT
  Arms: High concentration (370)
Procedure: CT angiography with low concentration contrast agent (320) — Two interventional arms use two different low concentration of iodine contrast agents, which is 320mgI/ml and 270mgI/ml respectively.
  Arms: Low concentration (320)
Procedure: CT angiography with low concentration contrast agent (270) — Two interventional arms use two different low concentration of iodine contrast agents, which is 320mgI/ml and 270mgI/ml respectively.
  Arms: Low concentration (270)

SUMMARY:
According to CT technology development, cardiac CT is very useful examination as noninvasive examination and the accuracy in locating lesions has increased to 95%. Specifically, cardiac CT has been performing a gateway role in reducing invasive cardiac angiography implemented solely for the purpose of diagnosis because of the invasive testing of makeshift cardiac angiography. However, cardiac CT also comes with the disadvantage that patients cannot avoid being exposed to radiation, so there has been much effort in appealing to reduce exposed radiation dose. Of these methods, the most effective is the method of repeatedly reconstitution by way of synchronized prospective ECG while using low tube-based potential. According to recent studies, the SNR(Signal Noise Ratio) and CNR(Contrast Noise Ratio) values representing image quality have been higher compared to the combined method of image reconstruction by makeshift filtered back projection and condition of image acquisition by patient BMI. Also, the administered amount of contrast agent can be reduced for achieving the same contrast effect due to the advantage of the increased effect of contrast enhancement by using low tube voltage. Therefore, the efficacy studies of using low concentration of contrast agents in conditions of using low tube voltage are being processed.

This study intends to prove that image quality does not deteriorate by suitable image reconstruction method with low concentration contrast agent compared to the combined method of the makeshift filtered back projection image reconstruction method and the conditions of image acquisition according to BMI with general amount of contrast agent.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 20 years old
* Subject who had requested a coronary CT angiography as per a clinical disease

Exclusion Criteria:

* Subject suspected as having myocardial infarction, unstable angina pectoris, coronary artery disease
* Subject with heart attack within 40 days prior to the CT scan
* Subject with diagnosed complicated heart anomaly
* BMI (body mass index) > 35kg/m2
* Serum creatinine ≥1.5mg/dl of renal insufficiency
* Subject with pregnancy or unknown pregnancy
* Subject with history of hypersensitivity reaction of contrast agents
* Subject has contraindication of using nitroglycerine
* Subject has plan to participate or enrolled in other randomized clinical trial for cardiovascular disease.
* Subject has contraindication of using adenosine (e.g. bronchial asthma, 2-3 degree AV block, sick sinus syndrome, SBP (systolic blood pressure) less than 90mmHg, recent prescribed history of dipyridamole, hypersensitivity of adenosine)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07-10; Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Assess HU (Hounsfield unit) for image quality of 3 different protocol of contrast media in coronary CT angiography | 7 days

SECONDARY OUTCOMES:
Qualitative evaluation of image quality of coronary artery | 7 days
  Measurement of evaluable segment with 4 point grading system as visual assessment
Quantitative analysis of image quality using measuring HU | 7 days
  Measurement of HU (Hounsfield unit) of myocardium during adenosine stress test in static perfusion CT
Diagnostic accuracy of coronary CT angiography compared to invasive coronary angiography | 7 days
  On segment-basis analysis, sensitivity, specificity, positive negative predictive value, negative predictive value, and accuracy of CT angiography for diagnosis of presence of CAD which is defined by more than 50% diameter stenosis compared to invasive coronary angiography, will be calculated and compared between different concentration of contrast agents by means of generalized estimating equation based on binary logistic model.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Im DJ, Kim YH, Choo KS, Kang JW, Jung JI, Won Y, Kim HR, Chung MH, Han K, Choi BW. Comparison of coronary computed tomography angiography image quality with high- and low-concentration contrast agents (CONCENTRATE): study protocol for a randomized controlled trial. Trials. 2016 Jul 15;17(1):315. doi: 10.1186/s13063-016-1441-y. PMID 27418333